CLINICAL TRIAL: NCT06157229
Title: Multifactorial Approach Training for Anterior Shoulder Instability in Patients Undergoing Arthroscopic Bankart Repair, a Randomized Controlled Trial
Brief Title: Multifactorial Approach Training for Anterior Shoulder Instability in Patients Undergoing Arthroscopic Bankart Repair
Acronym: MATASI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spaarne Gasthuis (Other)
Collaborators: OLVG (Network); Ziekenhuis Amstelland (Other); Gelre Hospitals (Other); Medisch Spectrum Twente (Other); Flevoziekenhuis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: reudctionapprehension
Record Dates: First submitted 2023-06-20; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Shoulder Instability; Shoulder Dislocation or Subluxation; Fear of Movement; Kinesiophobia
MeSH Terms: conditions — Shoulder Dislocation; Joint Dislocations; Kinesiophobia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multifactorial Approach Training (MAT) (Experimental): MAT involves an evidence-based core outcome-set of interventions aimed at both regaining functional stability of the shoulder and also diminishing fear of (recurrent) dislocation and kinesiophobia. The protocol is based on a recent international Delphi-based consensus study, initiated since no protocol yet existed focusing on this psychological component of traumatic anterior shoulder instability.
  Interventions: Other: MAT
- Conventional Arthroscopic Bankart Repair Rehabilitation (CABRR) (Active Comparator): The original guidelines which most physiotherapists use throughout the rehabilitation of their patients following ABR is the ASSET guideline [2].
  Interventions: Other: CABRR

INTERVENTIONS:
Other: MAT — The protocol consists of four phases: 1) immobilization phase, 2) early protective phase, 3) intermediate phase and 4) late phase. The detailed guideline can be found in the following article:
  Gaunt, B. W., Shaffer, M. A., Sauers, E. L., Michener, L. A., McCluskey, G. M., & Thigpen, C. A. (2010). The American Society of Shoulder and Elbow Therapists' Consensus Rehabilitation Guideline for Arthroscopic Anterior Capsulolabral Repair of the Shoulder. Journal of Orthopaedic & Sports Physical Therapy, 40(3), 155-168. https://doi.org/10.2519/jospt.2010.3186
  Arms: Multifactorial Approach Training (MAT)
Other: CABRR — The protocol consists of four phases: 1) immobilization phase, 2) early phase, 3) intermediate phase and 4) advanced phase.
  The protocol comprises education, modified cognitive behavioral therapy, neuromuscular control exercises, kinetic chain exercises, range of motion enhancing exercises, strength and conditioning exercises, and sport-specific exercises. The protocol is currently unpublished.
  Arms: Conventional Arthroscopic Bankart Repair Rehabilitation (CABRR)

SUMMARY:
This study will compare functional outcomes after an arthroscopic Bankart repair between patients that underwent conventional arthroscopic Bankart repair rehabilitation, following the American Society of Shoulder and Elbow Therapists guideline and patients that underwent 'multifactorial approach training', which focusses on decreasing kinesiophobia and fear of recurrent dislocations.

The study population comprises patients who will undergo Arthroscopic Bankart Repair (ABR) after a traumatic anterior shoulder dislocation at Spaarne Gasthuis Haarlem/Hoofddorp, OLVG Amsterdam, Amstelland Ziekenhuis Amstelveen, Gelre Ziekenhuizen, Medisch Spectrum Twente, or Flevoziekenhuis Almere.

DETAILED DESCRIPTION:
Background: Fear for (recurrent) dislocation is a frequently reported patient perception regarding the treatment of anterior shoulder instability and is associated with poor outcomes like decrease in quality of life and unsuccesful return to sport. There is lack of standard multifactorial aftercare of shoulder instability surgery incorporating the psychological component of the experiences trauma of patients with shoulder instability. Therefore, a newly developed Rehabilitation Protocol (REPRO) aims to reduce fear for dislocation in order to increase psychological readiness to return to sport. The aim of this study is to compare the effect on the psychological readiness to return to sport between our new Multifactorial Approach Training (MAT) and Conventional Arthroscopic Bankart Repair Rehabilitation (CABRR) in a single-blinded, multi-center randomized controlled trial.

Methods: Patients, aged 18-67 years, with traumatic anterior shoulder instability, undergoing ABR will be included. Rehabilitation is started within 4 weeks following surgical treatment. Patients will be randomized to either the control group (A) or the MAT group (B). Group A will receive CABRR, according to the American Society of Shoulder and Elbow Therapists (ASSET) guidelines. Group B will receive MAT, following the REPRO. A total of 92 patients will be included, with 46 patients per study arm. Patients will be followed-up for 52 weeks. The primary outcome is change from baseline (surgical intervention; ABR) in Shoulder Instability Return to Sport Index (SIRSI) at 26 weeks postoperatively. Secondary outcomes include Oxford Shoulder Instability Score (OSIS), Subjective Shoulder Value (SSV), fear for dislocation measured with a Numeric Rating Scale (NRS), Tampa Scale of Kinesiophobia in patients with Shoulder Instability (TSK-SI), World Health Organization Quality of Life Questionnaire - BREF (WHOQoL-BREF), Return To Work (RTW), Return To Sports (RTS), shoulder pain measured with a NRS, , number of physiotherapy and outpatient clinic visits and patient satisfaction (VAS). At baseline and at 26 weeks postoperatively patients will undergo a task-based brain activity analysis using functional Magnetic Resonance Imaging (fMRI) to determine functional cerebral changes after treatment. The MATASI trial is to be conducted between 2024 and 2026.

ELIGIBILITY:
Inclusion Criteria:

* Primary or recurrent traumatic anterior shoulder dislocation (MRI-confirmed labral tear)
* Aged between 18-67 years
* Planned arthroscopic Bankart repair (ABR) surgery
* Understanding of spoken and written Dutch language
* Written informed consent (according to the ICH-GCP guidelines)
* Positive apprehension sign at physical examination

Exclusion Criteria:

* Posterior or multidirectional shoulder instability
* Presence of hyperlaxity of the upper extremity and absence of sulcus sign and >85 degrees of external rotation with the arm at the side at physical examination
* Connective tissue disorders (e.g. Ehlers-Danlos)
* Aged <18 or >67 years
* Assymetry in rotator cuff strength, bilateral component ((sub)luxations on contralateral side)
* History of soft tissue repair or bone block procedure on one of both shoulders
* Current or past anxiety disorders or use of anxiety supressing drugs (e.g. anti-psychotics)
* Implantable cardioverter defibrillator (ICD) (unable to be included for functional MRI)
* Neurological disorders or systemic disease
* Loss of anteroinferior sclerotic contour of the glenoid on AP view of the shoulder
* Hill-Sachs lesion visible on external rotation radiographs
* Greater tubercle fracture

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Shoulder Instability Return to Sport Index (SIRSI) | 26 weeks postoperative
  Patient reported outcome measure to assess psychological readiness to return to sport in patients with shoulder instability

SECONDARY OUTCOMES:
Oxford Shoulder Instability Score (OSIS) | 26 and 52 weeks postoperative
  Patient reported shoulder function between MAT and CABRR
Shoulder function, measured by Subjective Shoulder value (SSV) | baseline, 26 and 52 weeks postoperative
  Shoulder function, measured by Subjective Shoulder value (SSV)
Fear of recurrent dislocation, measured by Numeric Rating Scale (NRS) | baseline, 26 and 52 weeks postoperative
  Fear of recurrent dislocation, measured by Numeric Rating Scale (NRS)
Tampa Scale for Kinesiophobia in patients with Shoulder Instability (TSK-SI) | baseline, 26 and 52 weeks postoperative
  Patient reported outcome measure to assess the degree of kinesiophobia
World Health Organization Qualitiy of Life Questionnaire - BREF (WHOQoL-BREF) | baseline, 26 and 52 weeks postoperative
  Patient reported outcome measure to assess the self reported quality of life
Level of shoulder pain measured by Visual Analogue Scale (VAS) | baseline, 26 and 52 weeks postoperative
  Level of shoulder pain measured by Visual Analogue Scale (VAS)
Number of patients that return to work (RTW) following the surgery | 26 and 52 weeks postoperative
  Number of patients that return to work (RTW) following the surgery
Number of patients tha return to sport (RTS) following the surgery | 26 and 52 weeks postoperative
  Number of patients tha return to sport (RTS) following the surgery
Patient satisfaction regarding the surgical treatment and rehabilitation, measured by VAS | baseline, 26 weeks and 52 weeks postoperative
  Patient satisfaction regarding the surgical treatment and rehabilitation, measured by VAS
The number of physiotherapy and orthopedic surgeon visits | From start to end of treatment
  The number of physiotherapy and orthopedic surgeon visits
Task-based brain activity, measured in voxels | baseline and 26 weeks postoperative
  Analysis using functional Magnetic Resonance Imaging (fMRI) to determine functional cerebral changes after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Arthur van Noort, MD PhD, Principal Investigator — Orthopedic Surgeon and Head of Residency Program, Spaarne Gasthuis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaunt BW, Shaffer MA, Sauers EL, Michener LA, McCluskey GM, Thigpen C; American Society of Shoulder and Elbow Therapists. The American Society of Shoulder and Elbow Therapists' consensus rehabilitation guideline for arthroscopic anterior capsulolabral repair of the shoulder. J Orthop Sports Phys Ther. 2010 Mar;40(3):155-68. doi: 10.2519/jospt.2010.3186. PMID 20195022
- [Background] van Iersel TP, Tutuhatunewa ED, Kaman I, Twigt BA, Vorrink SN, van den Bekerom MP, van Deurzen DF. Patient perceptions after the operative and nonoperative treatment of shoulder instability: A qualitative focus group study. Shoulder Elbow. 2023 Oct;15(5):497-504. doi: 10.1177/17585732221122363. Epub 2022 Aug 24. PMID 37811392